CLINICAL TRIAL: NCT04106245
Title: The Effect of an EHealth Coaching Program on Patient Reported Outcomes of Men With Prostate Cancer
Brief Title: Effect of EHealth Coaching Program on Patient Reported Outcomes of Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0422; NCI-2019-05856 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0422 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (PACK health coach, survey) (Experimental): Patients are contacted once weekly by a health coach by text message, phone call, email, or a mobile application, for 3 months. The total time interacting with the health coach is about 3.5-4.5 hours across the study. Patients also complete surveys over 30 minutes each time at baseline and every 30 days for 3 months.
  Interventions: Behavioral: Behavioral Intervention; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Participate in PACK Health
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Survey Administration — Complete survey

SUMMARY:
This trial studies the effect of an eHealth coaching program (PACK Health) on patient reported outcomes of men with prostate cancer. An electronic health support program may affect prostate cancer patients' reported side effects and outcomes of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To model the trajectory of patient reported outcomes (PROs), as measured by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale (version [v]1.2), among men newly diagnosed with prostate cancer who are engaged in either active surveillance or active treatment, while enrolled in an e-health coaching program.

Ia. To compare the trajectories of (PROs) between men who are engaged in either active surveillance or active treatment, while enrolled in an e-health coaching program.

SECONDARY OBJECTIVES:

I. To evaluate the effect of digital health coaching program on:

Ia. Physical and mental health of men newly diagnosed with prostate cancer as measured by the subscales of the PROMIS Global Health Scale (v 1.2).

Ib. The global health outcomes of men with prostate cancer who are in active treatment by active treatment type (i.e. surgery, radiation, chemotherapy, hormonal therapy, or a combination of these methodologies).

Ic. The symptom experience of men newly diagnosed with prostate cancer as measured by the MD Anderson Symptom Inventory (MDASI).

Id. The frequency of emergency room visits and hospital admissions for patients receiving treatment in the ambulatory setting.

II. To evaluate the relationship between financial toxicity, as measured by the Consumer Score for Financial Toxicity (COST), and quality of life, as measured by the Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP).

OUTLINE:

Patients are contacted once weekly by a health coach by text message, phone call, email, or a mobile application, for 3 months. The total time interacting with the health coach is about 3.5-4.5 hours across the study. Patients also complete surveys over 30 minutes each time at baseline and every 30 days for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, speak and consent in English
* Newly diagnosed (within 6 months of diagnosis) with prostate cancer
* Internet access via smart phone, tablet, a computer, or another device with the capacity to receive calls, texts, or e-mails, as well as the electronic study assessments

Exclusion Criteria:

* Individuals who are terminally ill, defined as individuals identified by their physician as likely having 6 months or less to live, or those individuals transitioned to hospice care
* Individuals who have a prior diagnosis of prostate cancer
* Individuals for whom there is documentation of inability to provide consent in the medical record

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Model trajectories of men who participate in eHealth program | Up to 3 months
  Summary statistics and box plots will also be used to describe Patient Reported Outcomes Measurement Information System (PROMIS) (1.2) and other inventory scores and subscale scores by cohort and assessment time. A linear mixed effects model will be used to assess PROMIS (version 1.2) (and scores over time). The models will include assessment time, treatment and a treatment by time interaction as fixed effects and intercept as a random effect.
The number of emergency room visits | Baseline through day 90
  A generalized linear mixed model (GLMM) using a log link function will be used to model the number of emergency room visits. Generalized linear mixed Tobit models will be used if the data are found to be zero-inflated.
Number of hospital admissions | Baseline through day 90
  A GLMM using a log link function will be used to model the number of emergency room visits. Generalized linear mixed Tobit models will be used if the data are found to be zero-inflated.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Hacker, BS,PHD,RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org